CLINICAL TRIAL: NCT00284440
Title: Relationship Between Visual Field Progression in Glaucoma and Choroidal Blood Flow Response to the Hand-grip Test
Brief Title: Choroidal Blood Flow Response to Hand-grip Test in Progressive Glaucoma
Status: Withdrawn | Type: Observational
Why Stopped: enrollment problems
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 072-Leh-2005-001
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Visual field progression; Choroidal blood flow
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study is designed to compare the response of choroidal blood flow to the hand-grip test in glaucoma patients with and without visual field progression.

DETAILED DESCRIPTION:
Glaucoma is a worldwide leading cause of blindness. The key features of glaucoma are damage to the optic nerve head and progressive visual field defect, which is not necessarily only related to an increase in intraocular pressure. It has been suggested that ocular blood flow alterations in glaucoma are related to systemic vascular dysregulations.The hand-grip test has been suggested as a potential tool to unravel vascular dysregulation in the ocular circulation. Although applied routinely in clinical practice, a proper study testing the effectiveness of this test is lacking. The present study is designed to compare the response of choroidal blood flow to the hand-grip test in glaucoma patients with and without visual field progression.

ELIGIBILITY:
Inclusion Criteria: Patients fulfilling two out of three of the following criteria in one or both eyes: a) typical glaucomatous disc, b) visual field damage (a cluster of three points (except rim points) in at least one hemifield reduced by 5 dB or greater and including at least one point reduced by 10 dB or greater; a cluster of two points reduced by 10 dB or greater; or three adjacent points on the nasal horizontal meridian that differed by 5 dB or greater from their mirror points on the opposite side of the meridian), c) intraocular pressure above 21 mm Hg at least at one occasion. Furthermore, patients need to have a series of at least 5 visual field examinations, after exclusion of the first test, for assessment of progression.

-

Exclusion Criteria:

* Ametropia > 3dpt
* Inadequate transparency of ocular media as defined by physical examination
* Iridocorneal angle extremely narrow with complete or partial closure as determined by gonioscopy
* Any abnormality which in the physician's view would prevent reliable applanation tonometry or LDF of at least one eye
* History of chronic or recurrent severe inflammatory eye disease such as scleritis or uveitis
* History of ocular trauma or intraocular surgery within the past 6 months
* History of infection or inflammation within the past 3 months
* History of clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy or retinal detachment
* Patients with a significant history and/or active alcohol or drug abuse (significant is defined as that which in the opinion of the investigator may either put the patient at risk because of participation in the study or may influence the results of the study or the patient's ability to participate in the study).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orguel, MD, Principal Investigator — Chief of department of diagnostics
Locations (1):
- University Eye Clinic, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Gugleta K, Orgul S, Hasler PW, Picornell T, Gherghel D, Flammer J. Choroidal vascular reaction to hand-grip stress in subjects with vasospasm and its relevance in glaucoma. Invest Ophthalmol Vis Sci. 2003 Apr;44(4):1573-80. doi: 10.1167/iovs.02-0521. PMID 12657594
- See also: University Eye Clinic Basel, Switzerland — http://www.unispital-basel.ch/augenklinik.php